CLINICAL TRIAL: NCT01223040
Title: An Open-Label, Single-Center Study Evaluating the Effect of Systane Balance on Video Ocular Protection Index (OPI) and Blink Patterns in Patients Diagnosed With Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-09-64
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SYSTANE® Balance Lubricant Eye Drops (Experimental): SYSTANE Balance Lubricant Eye Drops dosed (bilaterally) in the office during each visit. Between visits 2 and 3, patients will dose 4 times per day for the 7 day period.
  Interventions: Other: SYSTANE® Balance Lubricant Eye Drops

INTERVENTIONS:
Other: SYSTANE® Balance Lubricant Eye Drops — Subjects will be dosed (bilaterally) in the office during each visit. Between visits 2 and 3, patients will dose 4 times per day for the 7 day period.

SUMMARY:
The purpose of this study is to evaluate the effect of acute and repeat dosing of Systane Balance on Video Ocular Protection Index (OPI) and Blink Patterns in a population of dry eye patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have history of mild-moderate dry eye with use of (or desire to use) eye drops in past 6 months

Exclusion Criteria:

* Patients cannot wear contact lenses within 1 week prior nor during the study, and cannot have a history of hypersensitivity to any component of Systane Balance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Changes in video Ocular Protection Index 10 and 55 minutes following Systane Balance instillation at Days 1 and 7. | 8 days

SECONDARY OUTCOMES:
Changes in blink pattern in subjects with mean Interblink Interval (IBI) < 3 seconds at Days 2 and 8 | 9 days
Fluorescein staining at Visits 1 & 3 on the Ora staining scale | 9 days
Ocular Symptomology at each visit | 9 days